CLINICAL TRIAL: NCT02004379
Title: Register of Telaprevir and Boceprevir in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-TEL-2013-01
Record Dates: First submitted 2013-11-20; First posted 2013-12-09 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C; telaprevir; boceprevir; clinical practice
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with hepatitis C, genotype 1: Patients with hepatitis C, genotype 1, treated with telaprevir or boceprevir

SUMMARY:
Know through routine clinical practice the effectiveness and safety of current treatment of hepatitis C virus, genotype 1, for patients who have never been treated and for patients who have been previously treated

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by hepatitis C virus, genotype 1
* Indication of treatment with telaprevir or boceprevir in F3 and F4 fibrosis

Exclusion Criteria:

* Being taking part in other
* Inability to follow a monitoring
* Contra-indications on triple therapy
* Coinfected with HIV and HBV (hepatitis B virus)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis C, genotype 1, who are elegible to be treated with telaprevir or boceprevir
Sampling Method: Non-Probability Sample
Enrollment: 1553 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of current treatment of hepatitis C virus, genotype 1, for patients who have never been treated and for patients who have been previously treated | 12 months
  Know through routine clinical practice the percentage of patients who have negative VHC-ARN
Safety of current treatment of hepatitis C virus, genotype 1, for patients who have never been treated and for patients who have been previously treated | 12 months
  Number and frequencies of serious adverse event (SAE) during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Javier Salmerón Escobar, Principal Investigator — Hospital Universitario de San Cecilio
Locations (48):
- Spain (48):
  - Hospital Universitario Doctor Negrín, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Comarcal Santa Ana, Motril, Granada
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital General Universitario Rafael Méndez, Lorca, Murcia
  - Agencia Sanitaria Costa del Sol, Marbella, Málaga
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitario A Coruña, A Coruña
  - Hospital de Poniente, Almería
  - Hospital Torrecárdenas, Almería
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitario de San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital de Guadalajara, Guadalajara
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital San Jorge, Huesca
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital de León, León
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Morales Meseguer, Murcia
  - Hospital Reina Sofía, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Unviersitario Virgen del Rocío, Seville
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital General de Valencia, Valencia
  - Hospital la Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital de Zamora, Zamora
  - Hospital Clínico Universitario de Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Salmeron J, Vinaixa C, Berenguer R, Pascasio JM, Sanchez Ruano JJ, Serra MA, Gila A, Diago M, Romero-Gomez M, Navarro JM, Testillano M, Fernandez C, Espinosa D, Carmona I, Pons JA, Jorquera F, Rodriguez FJ, Perez R, Montero JL, Granados R, Fernandez M, Martin AB, Munoz de Rueda P, Quiles R; Alhambra Spanish Study Group. Effectiveness and safety of first-generation protease inhibitors in clinical practice: Hepatitis C virus patients with advanced fibrosis. World J Gastroenterol. 2015 Aug 14;21(30):9163-74. doi: 10.3748/wjg.v21.i30.9163. PMID 26290644